CLINICAL TRIAL: NCT02574182
Title: Walking, Brain and Functional Magnetic Resonance Imaging Study of Motor Representations in Healthy Subjects and Amnestic MCI
Brief Title: Study of Motor Representations in Healthy Subjects and Amnestic MCI
Acronym: IRMARCHE
Status: Completed | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: CHU PROMOTEUR 2014/32
Record Dates: First submitted 2015-09-18; First posted 2015-10-12 (Estimated); Last update posted 2021-07-12 (Actual); Status verified 2021-07

CONDITIONS: Mild Cognitive Impairment
Keywords: Mild Cognitive Impairment; Magnetic Resonance Imaging
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Control subjects under 40 years: Brain MRI Simulated walking with Corvit boots Records gait parameters on Gaitrite carpet
  Interventions: Radiation: Brain MRI
- Control subjects over 60 years: Brain MRI Simulated walking with Corvit boots Records gait parameters on Gaitrite carpet
  Interventions: Radiation: Brain MRI
- MCI subjects over 60 years: Brain MRI Simulated walking with Corvit boots Records gait parameters on Gaitrite carpet
  Interventions: Radiation: Brain MRI

INTERVENTIONS:
Radiation: Brain MRI — Brain MRI (Magnetic Resonance Imaging) brain is a painless test that allows to visualize the different brain structures.
  Korvit, device made up of 2 shoes which reproduces the feeling to go. The Korvit® system appears possible to analyze the activated cerebral zones and to thus try to better understand the operation of the brain during walk.
  The GAITRite is a carpet for recording the walking operating parameters
  Other Names: KORVIT; GAITRite

SUMMARY:
Walking, Brain and Functional Magnetic Resonance Imaging Study of motor representations in healthy subjects and amnesic MCI.

DETAILED DESCRIPTION:
Review and compare mapping brain activation in Magnetic Resonance Imaging about healthy subjects according to age (<40 years and> 60 years) and MCI through the combination of two paradigms: on mechanically simulated by Korvit® boots and imagination of the walk.

ELIGIBILITY:
Inclusion Criteria:

* Obtaining the signature of consent to participation in the study
* Age above 18 years
* Lack dementia as NICDS-ADRDA criteria
* Lack of pre-existing musculoskeletal disorders, regardless of the cause (except MCI).
* Absence of a history of stroke or other cerebrovascular disease with spinal sensorimotor sequelae.
* No cons-indication for performing a brain MRI.
* Witennses, population of young (<40 years)
* Witnesses ,population of older subjects (> 60 years)
* Witnesses Lack of MCI
* MCI patients, criteria MCI criteria according to Dubois

Exclusion Criteria :

* Refusal of MRI.
* Contraindications to brain MRI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Healthy volunteers over 18 and under 40.
  * Healthy volunteers over 60 years.
  * MCI patient over 60 years
Sampling Method: Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2015-02-24 (Actual); Primary Completion 2017-05-13 (Actual); Study Completion 2017-05-13 (Actual)

PRIMARY OUTCOMES:
Review and compare mapping cerebral activation in brain MRI | One day
  Review and compare mapping brain activation in healthy about MRI according to age (<40 years and> 60 years) and MCI through the combination of two paradigms: on mechanically simulated by Korvit® boots and imagination the walk. The primary endpoint is the analysis of fMRI brain mapping in accordance with the different paradigms of acquisition. The MRI data will be the subject of a specific statistical treatment, via dedicated software, which will be implemented under the control of the investigators who have conducted such an fMRI analysis in previous studies. Various brain mapping can be established from the data collected. It may include statistical comparisons between different preselected regions, and different experimental conditions, or correlation studies between brain activation and clinical parameters.

SECONDARY OUTCOMES:
Review and compare mapping brain activation in healthy subjects and MCI MRI in imagination alone walking. | One day
  Review and compare mapping brain activation in healthy subjects and MCI MRI in imagination alone walking. the secondary endpoint will be the analysis of spatiotemporal gait parameters
Study of differences in terms of activation of brain mapping | One day
  Study of differences in terms of activation of brain mapping between mechanical stimulation task arch simulating the place of the step (pace to 120 steps per minute) and a random mechanical stimulation (not reproducing the place of the pitch) . the secondary endpoint will be the analysis of spatiotemporal gait parameters
study of functional connectivity of sensorimotor cortex obtained by fMRI resting in the subject MCI. | One day
  study of functional connectivity of sensorimotor cortex obtained by fMRI resting in the subject MCI. the secondary endpoint will be the analysis of spatiotemporal gait parameters
study of the potential effects on muscle activation, and autonomic nervous system | One day
  study of the potential effects on muscle activation, and autonomic nervous system of plantar mechanical stimulation reproducing walking. the secondary endpoint will be the analysis of spatiotemporal gait parameters

CONTACTS AND LOCATIONS:
Overall Officials: Michael Dinomais, MD, Principal Investigator — UH Angers
Locations (1):
- University Hospital Angers, Angers, Pays de la Loire Region, France

REFERENCES:
- [Background] Dinomais M, Minassian AT, Tuilier T, Delion M, Wilke M, N'Guyen S, Richard I, Aube C, Menei P. Functional MRI comparison of passive and active movement: possible inhibitory role of supplementary motor area. Neuroreport. 2009 Oct 7;20(15):1351-5. doi: 10.1097/WNR.0b013e328330cd43. PMID 19734813
- [Background] Beauchet O, Allali G, Berrut G, Hommet C, Dubost V, Assal F. Gait analysis in demented subjects: Interests and perspectives. Neuropsychiatr Dis Treat. 2008 Feb;4(1):155-60. doi: 10.2147/ndt.s2070. PMID 18728766
- [Background] Rimmer E, Wojciechowska M, Stave C, Sganga A, O'Connell B. Implications of the Facing Dementia Survey for the general population, patients and caregivers across Europe. Int J Clin Pract Suppl. 2005 Mar;(146):17-24. doi: 10.1111/j.1368-504x.2005.00482.x. PMID 15801187
- [Background] Ogawa S, Lee TM, Nayak AS, Glynn P. Oxygenation-sensitive contrast in magnetic resonance image of rodent brain at high magnetic fields. Magn Reson Med. 1990 Apr;14(1):68-78. doi: 10.1002/mrm.1910140108. PMID 2161986
- [Background] Beauchet O, Allali G, Launay C, Herrmann FR, Annweiler C. Gait variability at fast-pace walking speed: a biomarker of mild cognitive impairment? J Nutr Health Aging. 2013 Mar;17(3):235-9. doi: 10.1007/s12603-012-0394-4. PMID 23459976